CLINICAL TRIAL: NCT07091357
Title: A Multicenter, Randomized, Double-blind, Placebo-controlled Phase II Clinical Study to Evaluate the Efficacy, Safety, Pharmacokinetics and Pharmacodynamics of SHR-1819 Injection in Patients With Seasonal Allergic Rhinitis
Brief Title: A Clinical Study on the Efficacy, Safety, Pharmacokinetics and Pharmacodynamics of SHR-1819 Injection in Patients With Seasonal Allergic Rhinitis
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Guangdong Hengrui Pharmaceutical Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SHR-1819-206
Record Dates: First submitted 2025-07-21; First posted 2025-07-29 (Actual); Last update posted 2025-09-03 (Actual); Status verified 2025-07

CONDITIONS: Seasonal Allergic Rhinitis
MeSH Terms: conditions — Rhinitis, Allergic, Seasonal

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- SHR-1819 Injection Dose 1 Group (Experimental)
  Interventions: Drug: SHR-1819 Injection
- SHR-1819 Injection Dose 2 Group (Experimental)
  Interventions: Drug: SHR-1819 Injection
- SHR-1819 Injection Placebo Group (Placebo Comparator)
  Interventions: Drug: SHR-1819 Injection Placebo

INTERVENTIONS:
Drug: SHR-1819 Injection — SHR-1819 injection.
  Arms: SHR-1819 Injection Dose 1 Group; SHR-1819 Injection Dose 2 Group
Drug: SHR-1819 Injection Placebo — SHR-1819 injection placebo.
  Arms: SHR-1819 Injection Placebo Group

SUMMARY:
This is a trial to evaluate the safety and efficacy of SHR-1819 injection in the treatment of patients with seasonal allergic rhinitis.

ELIGIBILITY:
Inclusion Criteria:

1. At the time of signing the informed consent form, the age is 18 to 75 years old.
2. Meet the diagnostic criteria for seasonal allergic rhinitis (SAR) as defined in the Chinese Guidelines for the Diagnosis and Treatment of Allergic Rhinitis (2022, Revised Edition), with or without allergic conjunctivitis, and have a disease duration of at least 2 years.
3. At the screening visit, the investigator assesses that the subject had poor efficacy with intranasal glucocorticoids and/or other medications for allergic rhinitis (antihistamines, leukotriene receptor antagonists, etc.) during the same pollen season in the past.
4. The subject has an immunoglobulin E (IgE)-mediated hypersensitivity to at least one pollen allergen in the current season or the same period, which can be confirmed based on the skin prick test (SPT) and/or serum specific IgE results during the screening period (test results within 1 year before randomization are acceptable).
5. Willing and able to complete the patient diary as required by the protocol during the study period.
6. Female subjects of childbearing potential and male subjects whose partners are females of childbearing potential agree to use the contraceptive measures specified in the protocol from the signing of the ICF until 3 months after the last administration.

Exclusion Criteria:

1. During screening or within 2 weeks prior to the screening visit, the subject has other active rhinitis excluding SAR, including but not limited to infectious rhinitis, drug-induced rhinitis, vasomotor rhinitis, non-allergic rhinitis with eosinophilia syndrome, dry rhinitis, atrophic rhinitis, etc.
2. During screening or within 2 weeks prior to the screening visit, there may be other nasal comorbidities or concurrent diseases/states that could affect the judgment of efficacy (including but not limited to nasal polyps, cerebrospinal fluid rhinorrhea, severe nasal septal deviation, status after nasal or sinus surgery within 1 year, etc.), acute/chronic sinusitis (except those deemed non-influential by the investigator), or upper respiratory tract infections.
3. During screening, there is glaucoma, cataract, ocular simple herpes, other ocular infections such as infectious conjunctivitis, acute conjunctivitis, acute keratitis (except for symptoms related to allergic rhinitis).
4. During the screening visit, subjects with perennial allergic rhinitis (PAR) allergic to pet hair are included; if the subject currently has no contact with pet hair, they can be enrolled.
5. Subjects with severe asthma who are receiving treatment with inhaled glucocorticoids (ICS) at a daily high dose or equivalent of more than twice the standard dose.
6. Subjects who initiated ICS treatment for asthma within 4 weeks prior to the screening visit. If the subject has been treated with a stable dose of ICS for at least 4 weeks before the screening visit, and the ICS dosage does not exceed twice the daily high dose, and the investigator assesses that the asthma remains well-controlled during the study while maintaining this dosage, such subjects may be screened.
7. Within 3 months prior to the screening visit, the subject had an acute exacerbation of asthma requiring hospitalization for more than 24 hours.
8. Within 6 months prior to the screening visit, the subject has a history of vernal keratoconjunctivitis (VKC) and/or atopic keratoconjunctivitis (AKC).
9. Within 1 week prior to randomization, the subject has received treatment with the following medications: leukotriene receptor antagonists. If the subject has been stably using mast cell membrane stabilizers, decongestants, nasal anticholinergic drugs, or other nasal preparations that may affect SAR assessment for ≥1 week at the time of screening, they may be included.
10. Within 2 weeks prior to the screening visit, the subject has used monoamine oxidase inhibitors.
11. Within 4 weeks prior to the screening visit, the subject has received the following treatments: systemic glucocorticoids, systemic immunosuppressants (including but not limited to hydroxychloroquine, cyclosporine, azathioprine, methotrexate, cyclophosphamide, tacrolimus, etc.), systemic traditional Chinese medicines (including proprietary Chinese medicines) for treating allergic rhinitis, and tricyclic antidepressants.
12. Within 4 weeks prior to the screening visit, the subject initiated immunotherapy or plans to receive immunotherapy during the study. If the subject has maintained a stable dose of immunotherapy for 4 weeks before screening and can continue this dose throughout the study, they may be enrolled.
13. Within 8 weeks prior to the screening visit or within 5 half-lives (if the half-life is known) of receiving investigational drugs or medical devices, whichever is longer. If the subject participated in a clinical study but only signed the informed consent form, and it can be proven that screening failed and no medication was administered, they may be enrolled.
14. Within 3 months prior to the screening visit, the subject has received or been exposed to other live vaccines or live attenuated vaccines, or participated in a vaccine clinical trial.
15. Within 6 months prior to the screening visit, the subject has used other biological agents.
16. Within 1 week prior to the screening visit, the subject requires systemic antimicrobial treatment (for viral, bacterial, fungal, or parasitic infections).
17. At the time of screening and within 2 weeks prior to screening, positive results for human immunodeficiency virus antibody (HIV), syphilis antibody, and hepatitis C virus (HCV) antibody; hepatitis B virus (HBV) infection meets the following (test results within 2 weeks prior to screening are acceptable).
18. Within 3 months prior to the screening visit, the subject has undergone major surgery, or plans to undergo major surgery during the study period.
19. Within 6 months prior to the screening visit, the subject was diagnosed with active tuberculosis.
20. Within 6 months prior to the screening visit, the subject was diagnosed with or the investigator determined the presence of suspected immunosuppressive diseases.
21. Within 1 year prior to the screening visit, the subject has a history of recurrent herpes zoster or Kaposi varicelliform eruption (≥2 times), disseminated herpes zoster, or disseminated herpes simplex.
22. Has or has a history of malignant tumor (except for cutaneous squamous cell carcinoma, basal cell carcinoma, or cervical in situ carcinoma that has been completely resected and shows no evidence of recurrence).
23. Accompanied by other severe or chronic diseases that are poorly controlled.
24. Pregnant or lactating women.
25. Within 6 months prior to screening, the subject has a history of alcohol abuse.
26. The investigator determines that there are conditions affecting the safety and efficacy evaluation of the study drug, as well as any other circumstances that may lead to the patient's non-compliance with the trial procedures and log filling.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-08-06 (Actual); Primary Completion 2025-10 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
The mean change from baseline in daily retrospective total nasal symptom score (rTNSS). | Within 2 weeks of treatment.

SECONDARY OUTCOMES:
The mean change from baseline in daily retrospective total nasal symptom score (rTNSS). | Within 4 weeks of treatment.
The mean change rate from baseline in daily retrospective total nasal symptom score (rTNSS). | Within 2 weeks of treatment.
The mean change rate from baseline in daily retrospective total nasal symptom score (rTNSS). | Within 4 weeks of treatment.
Adverse events (AEs). | 12 weeks.

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Tongren Hospital, Capital Medical University, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided